CLINICAL TRIAL: NCT06305403
Title: Comparison of Venous Excess Ultrasound Score (VExUS) With Neutrophil Gelatinase-associated Lipocalin (NGAL) in the Diagnosis and Prognosis of Sepsis-associated Acute Kidney Injury
Brief Title: VEXUS and NGAL in the Diagnosis and Prognosis of Sepsis-associated Acute Kidney Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ayse Belin Ozer, Head of Intensive Care Unit, Inonu University
Other Study IDs: VEXUS1
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Sepsis; Acute Kidney Injury
Keywords: ngal; vexus
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples Without DNA — blood sample for blood ngal level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with sepsis who develop AKI
  Interventions: Diagnostic Test: serum creatinin level
- 2: Patients with sepsis who not develop AKI
  Interventions: Diagnostic Test: serum creatinin level

INTERVENTIONS:
Diagnostic Test: serum creatinin level — Serum creatinine and urine amounts will be checked for five days.
  Other Names: urine output

SUMMARY:
In this prospective observational study, patients hospitalized in mixed intensive care unit, aged between 18 and 80, and diagnosed with sepsis and septic shock according to sepsis-3 criteria will be included.

To determine whether patients develop AKI during the first five days of ICU admission, creatinine and urine output will be monitored daily for the first five days of ICU admission according to KDIGO criteria. Clinical diagnosis and treatment of AKI will be made according to KDIGO.

According to KDIGO, patients will be divided into two groups: those who develop AKI and those who do not.

By comparing plasma NGAL and VEXUS scores between groups, the sensitivity and specificity of the VEXUS score in determining AKI will be determined.

DETAILED DESCRIPTION:
In this prospective observational study, patients hospitalized in mixed intensive care unit, aged between 18 and 80, and diagnosed with sepsis and septic shock according to sepsis-3 criteria will be included.

Poor abdominal echogenicity, age < 18 years, other conditions causing shock (hypovolemic, cardiogenic, neurogenic), life expectancy less than 24 hours, pregnancy, vasospastic disease, intraperitoneal pressure > 15 mm Hg, obstructive renal failure or suspected renal artery Defined as the presence of stenosis, liver and kidney transplanted patients, liver and kidney tumors, patients receiving dialysis treatment, single kidney and other kidney abnormalities, right heart failure, acute mesenteric ischemia (GFR) < 30 ml/min/1.73m2. Those with severe acute or chronic renal failure will be excluded from the study.

After patients are diagnosed with sepsis/septic shock, in accordance with the Surviving Sepsis 2021 guide; Cultures will be sent and antibiotics, fluids, and vasopressor treatment will be started if necessary. Standard monitoring of the patients (heart rate, mean arterial pressure, peripheral oxygen saturation) will be performed.

To determine whether patients develop AKI during the first five days of ICU admission, creatinine and urine output will be monitored daily for the first five days of ICU admission according to KDIGO criteria. Clinical diagnosis and treatment of ACI will be made according to KDIGO.

According to KDIGO, patients will be divided into two groups: those who develop ACI and those who do not.

By comparing plasma NGAL and VEXUS scores between groups, the sensitivity and specificity of the VEXUS score in determining ACI will be determined.

Blood samples for plasma NGAL level will be taken within the first 24 hours of sepsis diagnosis, after the patient has received one-hour bundle therapy and the patient has been stabilized. The VEXUS score will be measured simultaneously with ultrasound. Both parameters will be repeated after the 72nd hour.

VEXUS score measurement will be performed by an experienced practitioner with a transparietal 2-5 MHz curvi-linear probe (Ch5-2 ultrasound transducer, Siemens Healthineers ACUSON NX3) and the values and graphs will be saved to external memory.

For plasma NGAL level, approximately 10 ml of blood samples taken from the peripheral vein will be centrifuged at 1500 rpm for 5 minutes and stored at -80 °C.

Patients' age, gender, weight, height, body mass index, accompanying diseases (e.g., diabetes mellitus, hypertension, heart failure, COPD, cancer, anemia, poisonings, trauma), source and type of infection, procalcitonin, c-reactive protein (CRP), lactate, routine markers of circulation, central venous pressure, medications (diuretic, vasopressor, inotropic agent, antimicrobial, insulin, colloid, albumin use, blood and blood product transfusion), recent use of contrast material, fluid balance, renal replacement. The need for treatment, the need for mechanical ventilation treatment, the stage of the AKI group according to KDIGO, Acute Physiology and Chronic Health Evaluation (APACHE II) score, Sequential Organ Failure Assesment (SOFA) score, hospital stay and 28-day mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* sepsis septic shock

Exclusion Criteria:

* Poor abdominal echogenicity,
* other conditions causing shock (hypovolemic, cardiogenic, neurogenic),
* life expectancy less than 24 hours, pregnancy, vasospastic disease, intraperitoneal pressure > 15 mm Hg, obstructive renal failure liver and kidney transplanted patients, liver and kidney tumors, patients receiving dialysis treatment, single kidney and other kidney abnormalities, right heart failure, acute mesenteric ischemia chronic renal failure

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: sepsis and septic shock in ICU
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-03-18 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
ngal | first and fifth days
  neutrophil gelatinase-associated lipocalin
VEXUS | first and fifth days
  venous excess ultrasound score (If VCI diameter is < 2 cm, there is no congestion. If the VExUS score is 0, and you do not need to proceed further. If VCI>2, congestion is present. Further examination is necessary to determine the severity of congestion and VExUS scores 1-3.Each of the hepatic, portal and renal veins are subsequently examined and classified as normal, mildly congested, or severely congested. The VExUS system has four grades: Grade 0 represents no congestion in any organ, Grade 1 represents only mild congestive findings, Grade 2 represents severe congestive findings in only one organ, and Grade 3 represents severe congestive findings in at least two out of three organ systems.

SECONDARY OUTCOMES:
MORTALİTY | 28 days
  28 days mortality

IPD SHARING:
Plan to Share IPD: Undecided